CLINICAL TRIAL: NCT05328323
Title: Turkish Translation, Cross-Cultural Adaptation and Validation of the of the Physical Activity and Social Support Scale
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Büşra Aksan Sadıkoğlu, PT, MSc, Istanbul University - Cerrahpasa
Other Study IDs: IstanbulUC2022
Record Dates: First submitted 2022-04-08; First posted 2022-04-14 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Social Support, Physical Activity, Validation, Reliability
Keywords: social support; physical activity; validity; reliability
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire application — Participants will be asked to fill in the "Physical Activity and Social Support Scale (PASSS)" adapted into Turkish. Evaluations of the participants will be made in the form of an online survey via "Google Forms". "Multidimensional Scale of Perceived Social Support and International Physical Activity Questionnaire" will be used for construct validity of the scale, and SF-12 physical and mental component summary scores will be used for convergent and divergent validity. The questionnaire will be repeated every 7-14 days in order to perform the test-retest analysis of the questionnaire.

SUMMARY:
Investigation of the connection between physical activity and social support has gained importance in recent years and there is evidence in the literature showing a positive relationship between social support and physical activity. The aim of this study is to translate the 20-item Physical Activity and Social Support Scale (PASSS), which was developed by Golaszewski and Bartholomew in 2019 to evaluate social support for physical activity, into Turkish, to provide cultural adaptation, and to perform a reliability and validity study of the translated version of the scale in healthy adults. Within the scope of the inclusion criteria, 230 healthy young adult individuals between the ages of 18-35, who do physical activity at least twice a week, who do not have serious limitations that prevent participation in physical activity, and who voluntarily agree to participate in the study by signing their consent, will be recruited.

As a result of the study, it is aimed to bring a valid and reliable tool in Turkish to the literature in order to evaluate the importance of social support on physical activity.

DETAILED DESCRIPTION:
Investigation of the connection between physical activity and social support has gained importance in recent years and there is evidence in the literature showing a positive relationship between social support and physical activity. The aim of this study is to translate the 20-item Physical Activity and Social Support Scale (PASSS), which was developed by Golaszewski and Bartholomew in 2019 to evaluate social support for physical activity, into Turkish, to provide cultural adaptation, and to perform a reliability and validity study of the translated version of the scale in healthy adults. Within the scope of the inclusion criteria, 230 healthy young adult individuals between the ages of 18-35, who do physical activity at least twice a week, who do not have serious limitations that prevent participation in physical activity, and who voluntarily agree to participate in the study by signing their consent, will be recruited. The demographic information of the participants will be obtained with the sociodemographic data form prepared to record the demographic information of the participants, and then the participants will be asked to fill in the "Physical Activity and Social Support Scale" adapted into Turkish. Evaluations of the participants will be made in the form of an online survey via "Google Forms". "Multidimensional Scale of Perceived Social Support and International Physical Activity Questionnaire" will be used for construct validity of the scale, and SF-12 physical and mental component summary scores will be used for convergent and divergent validity. The survey will be repeated every 7-14 days in order to perform the test-retest analysis of the survey. As a result of the study, it is aimed to bring a valid and reliable tool in Turkish to the literature in order to evaluate the importance of social support on physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-35
* Individuals who do physical activity at least 2 days a week

Exclusion Criteria:

* Severe physical limitations that prevent physical activity
* Individuals with cognitive impairment

Ages: 18 Years to 35 Years | Sex: All
Age Groups: Adult
Study Population: Young adult individuals aged 18-35 who have physical activity at least 2 days a week will be included the study.
Sampling Method: Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Physical Activity and Social Support Scale (PASSS) | Baseline (First assessment)
  The questionnaire, which was developed to evaluate social support for physical activity, consists of 20 questions and provides the opportunity to evaluate social support for physical activity in various dimensions.

SECONDARY OUTCOMES:
Physical Activity and Social Support Scale (PASSS) | Within a 7-to-14-day period after the first assessment (Second assessment)
  The questionnaire, which was developed to evaluate social support for physical activity, consists of 20 questions and provides the opportunity to evaluate social support for physical activity in various dimensions.
Multidimensional Scale of Perceived Social Support (MSPSS) | Baseline (First assessment)
  MSPSS is a 12-item scale that measures the adequacy of social support. It consists of 3 subgroups that include items about family, friends and social support from a special person. It consists of 4 items for each group and each item is graded on a 7-item likert scale. A high total score indicates a high level of perceived social support.
International Physical Activity Questionnaire-Short Form (IPAQ-Short Form) | Baseline (First assessment)
  IPAQ is a global scale that allows to evaluate physical activity. The short version provides information on time spent walking, moderate-intensity, vigorous activity, and sedentary activity. In the outcome evaluation, the estimation of MET energy expenditure for each activity category and the weekly reported activity time are used to calculate total physical activity.
SF-12 | Baseline (First assessment)
  Physical component-12 score is obtained from general health, physical role, physical functionality and body pain sub-dimensions. Mental component-12 score is obtained from mental health, emotional role, social functionality and energy sub-dimensions.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided